CLINICAL TRIAL: NCT03855228
Title: Safety and Efficacy of Mometasone Furoate Nasal Spray With the Addition of Loratadine Versus Placebo in the Treatment of Seasonal Allergic Rhinitis (Study No. C94-145)
Brief Title: Safety and Efficacy of Mometasone Furoate Nasal Spray With the Addition of Loratadine Versus Placebo in Participants With Seasonal Allergic Rhinitis (C94-145)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C94-145; C94-145 (Other: Schering-Plough Corporation Protocol Number)
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Results first posted 2019-07-26 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate; Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MFNS 200 µg + Loratadine 10 mg (Experimental): Daily administration of 200 µg of MFNS plus oral dose of 10 mg loratadine tablet.
  Interventions: Drug: Mometasone furoate nasal spray (MFNS); Drug: Loratadine
- MFNS 200 µg (Active Comparator): Daily administration of 200 µg of MFNS plus oral placebo tablet.
  Interventions: Drug: Mometasone furoate nasal spray (MFNS); Drug: Placebo tablet
- Loratadine 10 mg (Active Comparator): Daily administration of oral dose of 10 mg loratadine tablet plus placebo nasal spray.
  Interventions: Drug: Loratadine; Drug: Placebo nasal spray
- Placebo (Placebo Comparator): Daily administration of placebo nasal spray plus oral placebo tablet.
  Interventions: Drug: Placebo nasal spray; Drug: Placebo tablet

INTERVENTIONS:
Drug: Mometasone furoate nasal spray (MFNS) — Daily dose of 200 µg of mometasone furoate administered as a nasal spray for 15 days.
  Other Names: SCH 32088; MK-0887; NASONEX®
  Arms: MFNS 200 µg; MFNS 200 µg + Loratadine 10 mg
Drug: Loratadine — Daily dose of 10 mg of loratadine administered as an oral tablet for 15 days.
  Other Names: Claritin®
  Arms: Loratadine 10 mg; MFNS 200 µg + Loratadine 10 mg
Drug: Placebo nasal spray — Daily dose of placebo administered as a nasal spray for 15 days.
  Arms: Loratadine 10 mg; Placebo
Drug: Placebo tablet — Daily dose of placebo administered as an oral tablet for 15 days.
  Arms: MFNS 200 µg; Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mometasone furoate nasal spray (MFNS) with the addition of loratadine vs MFNS alone, loratadine alone, or placebo, in the treatment of patients with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* 2-year history of seasonal allergic rhinitis
* Positive skin test response to a local seasonal allergen (current, or performed in investigator's office within the past year)
* Good health and free of any unstable, clinically significant disease, other than allergic rhinitis, that would interfere with the study schedule or evaluation of seasonal allergic rhinitis

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Women of childbearing potential who are not using an acceptable form of birth control
* Significant history of metabolic, cardiovascular, neurologic, hematologic, hepatic, gastrointestinal, cerebrovascular, respiratory, or renal disease, or any other disorder which, in the judgment of the investigator, could interfere with the study, or require treatment which might interfere with the study
* Use of any chronic medication which could affect the course of seasonal allergic rhinitis
* Asthma requiring chronic use of inhaled or systemic corticosteroids (inhaled bronchodilators are permitted for asthma treatment)
* Current or history of frequent, clinically significant sinusitis or chronic purulent postnasal drip
* Upper respiratory tract or sinus infection that requires antibiotic therapy within the previous 2 weeks, or a viral upper respiratory infection (URI) within the 7 days prior to Screening
* Dependence upon nasal, oral or ocular decongestants, or nasal topical antihistamines, in the opinion of the investigator
* Has rhinitis medicamentosa
* Evidence of clinically significant nasal candidiasis
* Investigational drug use within the previous 30 days
* Nasal structural abnormalities, including large nasal polyps and marked septal deviation, that significantly interfere with nasal air flow
* Immunotherapy (desensitization therapy), unless on a stable maintenance schedule for at least one month prior to the Screening visit
* History of multiple drug allergies, allergy to antihistamines or corticoids
* History of psychosis, antagonistic personality, poor motivation, hypochondriasis, or any other emotional or intellectual problems that are likely to limit the validity of consent to participate in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 1995-03-01 (Actual); Primary Completion 1995-08-07 (Actual); Study Completion 1995-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MFNS 200 μg + Loratadine 10 mg: Daily administration of 200 μg of Mometasone Furoate Nasal Spray (MFNS) plus oral dose of 10 mg loratadine tablet.
- MFNS 200 μg: Daily administration of 200 μg of MFNS plus oral placebo tablet.
Period: Overall Study
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Started | 169 | 176 | 182 | 177
Treated | 169 | 176 | 181 (1 participant immediately dropped out prior to starting study intervention.) | 176 (1 participant immediately dropped out prior to starting study intervention.)
Completed | 166 | 167 | 174 | 158
Not Completed | 3 | 9 | 8 | 19
Not completed — Adverse Event | 2 | 4 | 4 | 8
Not completed — Treatment Failure | 1 | 2 | 1 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 2 | 1
Not completed — Did Not Meet Entry Requirements | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Includes all randomized participants who received ≥1 dose of study treatment.
Groups:
- MFNS 200 μg + Loratadine 10 mg: Daily administration of 200 μg of MFNS plus oral dose of 10 mg loratadine tablet.
- Total: Total of all reporting groups
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo | Total
Number analyzed (Participants) | 169 | 176 | 181 | 176 | 702
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.6 (13.1) | 25.6 (13.2) | 25.2 (12.6) | 25.6 (13.3) | 25.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 89 | 91 | 85 | 350
  Male | 84 | 87 | 90 | 91 | 352
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 7 | 7 | 30
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 162 | 167 | 174 | 169 | 672
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 3 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 12 | 7 | 12 | 41
  White | 150 | 154 | 164 | 154 | 622
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 10 | 7 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Nasal Symptom Score (Assessed by Participant)
Description: Mean change from baseline (CFB), averaged over study days 1-15, is calculated for total nasal symptom scores assessed by participants. Participants scored 4 symptoms (rhinorrhea; nasal stuffiness; nasal itching; sneezing) in diaries on a scale from 0 (none) to 3 (severe). Scores sum to a total nasal symptom score (range: 0-12); higher values indicate greater severity. A decrease in symptom severity is reflected by a negative CFB.
  CFB is the 15-day average score minus baseline score. Scores were recorded twice daily, in morning (AM) and night (PM). Average AM/PM scores are first calculated separately, then averaged together to compute the 15-day average score. If diary entries were missing, an average AM or PM score was not calculated. If neither average AM nor PM score was calculated, total 15-day average score was not calculated. Baseline score is an average of the three AM and three PM scores preceding treatment.
Time Frame: Baseline and days 1 through 15 (average of 15 days of treatment)
Population: Includes randomized participants with ≥1 valid post-Baseline visit, no major protocol violations, and evaluable data for the days 1-15 average.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 166 | 175 | 165
Score on a scale
  Baseline | 7.9 (2.2) | 7.8 (2.2) | 7.9 (2.2) | 8.0 (2.1)
  Change From Baseline Days 1-15 | -3.0 (2.6) | -2.7 (2.5) | -1.9 (2.2) | -1.4 (2.2)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.36, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.02, ANOVA

2. Primary Outcome: Change From Baseline in Total Symptom Score (Assessed by Participant)
Description: Mean change from baseline (CFB), averaged over study days 1-15, is calculated for total symptom scores assessed by participants. Participants scored 8 symptoms (rhinorrhea; nasal stuffiness; nasal itching; sneezing; itching/burning eyes; tearing/watering eyes; eye redness; and ear/palate itching) in diaries on a scale from 0 (none) to 3 (severe). Scores sum to a total symptom score (range: 0-24); higher values indicate greater severity. A decrease in symptom severity is reflected by a negative CFB.
  CFB is the 15-day average score minus baseline score. Scores were recorded twice daily, in morning (AM) and night (PM). Average AM/PM scores are first calculated separately, then averaged together to compute the 15-day average score. If diary entries were missing, an average AM or PM score was not calculated. If neither average AM nor PM score was calculated, total 15-day average score was not calculated. Baseline score is an average of the three AM and three PM scores preceding treatment.
Time Frame: Baseline and days 1 through 15 (average of 15 days of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 166 | 175 | 165
Score on a scale
  Baseline | 14.3 (4.1) | 14.2 (4.4) | 14.4 (4.5) | 14.6 (4.3)
  Change From Baseline Days 1-15 | -5.4 (4.8) | -4.8 (4.7) | -3.8 (4.2) | -2.7 (4.2)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.35, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.03, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.02, ANOVA

3. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score on Day 15 (Assessed by Physician)
Description: The mean change from baseline on study day 15 was calculated for total nasal symptom scores assessed by physician. Total nasal symptom scores are a composite of the following: rhinorrhea, nasal stuffiness (congestion), nasal itching, and sneezing scores. Physician scored each symptom during study visit at baseline and study day 15, on a scale from 0 (none) to 3 (severe), totaling to a composite score from 0-12 where a higher value indicates greater severity.
  A negative change from baseline indicates a decrease in symptom severity.
Time Frame: Baseline and study day 15
Population: All randomized participants with: ≥1 valid post-Baseline visit; no major protocol violations; and who had an observation for the respective endpoint prior to either significant dose noncompliance, or onset of an adverse event that may have interfered with allergic rhinitis assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 164 | 172 | 162
Score on a scale
  Baseline | 8.7 (1.8) | 8.6 (1.8) | 8.6 (1.7) | 8.8 (1.8)
  Change From Baseline Day 15: number analyzed (Participants) | 160 | 159 | 167 | 154
  Change From Baseline Day 15 | -4.4 (3.1) | -4.2 (2.8) | -3.1 (2.8) | -2.8 (2.8)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.77, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.45, ANOVA

4. Secondary Outcome: Change From Baseline in Total Symptom Score on Day 15 (Assessed by Physician)
Description: The mean change from baseline on study day 15 was calculated for total symptom scores assessed by physician. Total symptom scores are a composite of the following: rhinorrhea, nasal stuffiness (congestion), nasal itching, sneezing, itching/burning eyes, tearing/watering eyes, redness of the eyes, and itching of the ears or palate scores. Physician scored each symptom during study visit at baseline and study day 15, on a scale from 0 (none) to 3 (severe), totaling to a composite score from 0-24 where a higher value indicates greater severity.
  A negative change from baseline indicates a decrease in symptom severity.
Time Frame: Baseline and study day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 164 | 172 | 162
Score on a scale
  Baseline | 15.9 (3.1) | 16.1 (3.4) | 15.9 (3.2) | 16.2 (3.5)
  Change From Baseline Day 15: number analyzed (Participants) | 160 | 159 | 167 | 154
  Change From Baseline Day 15 | -8.2 (5.3) | -8.0 (5.1) | -6.2 (5.1) | -5.4 (5.3)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.99, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.08, ANOVA

5. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score on Day 8 (Assessed by Physician)
Description: The mean change from baseline on study day 15 was calculated for total nasal symptom scores assessed by physician. Total nasal symptom scores are a composite of the following: rhinorrhea, nasal stuffiness (congestion), nasal itching, and sneezing scores. Physician scored each symptom during study visit at baseline and study day 8, on a scale from 0 (none) to 3 (severe), totaling to a composite score from 0-12 where a higher value indicates greater severity.
  A negative change from baseline indicates a decrease in symptom severity.
Time Frame: Baseline and study day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 164 | 172 | 162
Score on a scale
  Baseline | 8.7 (1.8) | 8.6 (1.8) | 8.6 (1.7) | 8.8 (1.8)
  Change From Baseline Day 8: number analyzed (Participants) | 165 | 163 | 172 | 162
  Change From Baseline Day 8 | -3.7 (3.1) | -3.6 (2.7) | -2.6 (2.6) | -2.2 (2.5)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.85, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.17, ANOVA

6. Secondary Outcome: Change From Baseline in Total Symptom Score on Day 8 (Assessed by Physician)
Description: The mean change from baseline on study day 8 was calculated for total symptom scores assessed by physician. Total symptom scores are a composite of the following: rhinorrhea, nasal stuffiness (congestion), nasal itching, sneezing, itching/burning eyes, tearing/watering eyes, redness of the eyes, and itching of the ears or palate scores. Physician scored each symptom during study visit at baseline and study day 8, on a scale from 0 (none) to 3 (severe), totaling to a composite score from 0-24 where a higher value indicates greater severity.
  A negative change from baseline indicates a decrease in symptom severity.
Time Frame: Baseline and study day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 164 | 172 | 162
Score on a scale
  Baseline | 15.9 (3.1) | 16.1 (3.4) | 15.9 (3.2) | 16.2 (3.5)
  Change From Baseline Day 8: number analyzed (Participants) | 165 | 163 | 172 | 162
  Change From Baseline Day 8 | -7.0 (5.4) | -6.9 (4.9) | -5.2 (4.6) | -4.6 (4.7)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.88, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.22, ANOVA

7. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis (SAR) on Day 15 (Assessed by Physician)
Description: The mean change from baseline on study day 15 was calculated for overall condition of rhinitis. Physicians scored participant rhinitis condition during study visit at baseline and study day 15, on a scale from 0 (none) to 3 (severe). A higher value indicates greater severity.
  A negative change from baseline indicates a decrease in symptom severity.
Time Frame: Baseline and study day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 164 | 172 | 162
Score on a scale
  Baseline | 2.3 (0.5) | 2.3 (0.5) | 2.3 (0.5) | 2.3 (0.5)
  Change From Baseline Day 15: number analyzed (Participants) | 160 | 159 | 167 | 154
  Change From Baseline Day 15 | -0.9 (0.7) | -0.9 (0.7) | -0.6 (0.8) | -0.6 (0.7)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.65, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.92, ANOVA

8. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis (SAR) on Day 8 (Assessed by Physician)
Description: The mean change from baseline on study day 8 was calculated for overall condition of rhinitis. Physicians scored participant rhinitis condition during study visit at baseline and study day 8, on a scale from 0 (none) to 3 (severe). A higher value indicates greater severity.
  A negative change from baseline indicates a decrease in symptom severity.
Time Frame: Baseline and study day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 164 | 172 | 162
Score on a scale
  Baseline | 2.3 (0.5) | 2.3 (0.5) | 2.3 (0.5) | 2.3 (0.5)
  Change From Baseline Day 8: number analyzed (Participants) | 165 | 163 | 172 | 162
  Change From Baseline Day 8 | -0.8 (0.8) | -0.7 (0.7) | -0.5 (0.7) | -0.5 (0.7)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.95, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; This analysis compares Change From Baseline values; Test type: Superiority; p = 0.58, ANOVA

9. Secondary Outcome: Response to Therapy on Day 15 (Assessed by Physician)
Description: Mean response to therapy based on the participant's status relative to baseline. Physician scored participant's response on a scale from 1 (complete relief) to 5 (treatment failure) during study visit on study day 15. A higher value indicates weaker response.
Time Frame: Study day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 160 | 159 | 167 | 154
Score on a scale | 2.8 (1.0) | 3.0 (1.0) | 3.4 (1.1) | 3.4 (1.1)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; Test type: Superiority; p = 0.29, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; Test type: Superiority; p = 0.80, ANOVA

10. Secondary Outcome: Response to Therapy on Day 8 (Assessed by Physician)
Description: Mean response to therapy based on the participant's status relative to baseline. Physician scored participant's response on a scale from 1 (complete relief) to 5 (treatment failure) during study visit on study day 8. A higher value indicates weaker response.
Time Frame: Study day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MFNS 200 μg + Loratadine 10 mg | MFNS 200 μg | Loratadine 10 mg | Placebo
Number analyzed (Participants) | 165 | 163 | 172 | 162
Score on a scale | 3.0 (1.1) | 3.1 (1.0) | 3.4 (0.9) | 3.6 (1.0)
Statistical Analysis 1: Comparison: MFNS 200 μg + Loratadine 10 mg vs MFNS 200 μg; Test type: Superiority; p = 0.41, ANOVA
Statistical Analysis 2: Comparison: MFNS 200 μg + Loratadine 10 mg vs Loratadine 10 mg; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: MFNS 200 μg + Loratadine 10 mg vs Placebo; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 4: Comparison: MFNS 200 μg vs Loratadine 10 mg; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 5: Comparison: MFNS 200 μg vs Placebo; Test type: Superiority; p < 0.01, ANOVA
Statistical Analysis 6: Comparison: Loratadine 10 mg vs Placebo; Test type: Superiority; p = 0.08, ANOVA

ADVERSE EVENTS:
Time Frame: Up to approximately 45 days.
Description: Analysis population includes all randomized participants with at least one post-Baseline evaluation. Adverse event (AE) preferred terms were converted from WHO-ART dictionary to the MedDRA version 12.0.
Groups:
- MFNS Pus Loratadine: Daily administration of 200 μg of MFNS plus oral dose of 10 mg loratadine tablet.
- MFNS 200: Daily administration of 200 μg of MFNS plus oral placebo tablet.
- Loratadine: Daily administration of oral dose of 10 mg loratadine tablet plus placebo nasal spray.
Arm/Group | MFNS Pus Loratadine | MFNS 200 | Loratadine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/176 | 0/181 | 0/176
Serious Adverse Events (participants affected / at risk) | 0/169 | 0/176 | 0/181 | 0/176
Other Adverse Events (participants affected / at risk) | 22/169 | 22/176 | 33/181 | 21/176
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MFNS Pus Loratadine (N=169) | MFNS 200 (N=176) | Loratadine (N=181) | Placebo (N=176)
HEADACHE (Nervous system disorders) | 22 (35) | 22 (28) | 33 (41) | 21 (31)

LIMITATIONS AND CAVEATS:
AE Preferred Terms were converted from WHO-ART dictionary to the MedDRA version 12.0.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator agrees not to publish or publicly present any interim results of the Protocol study without the prior written consent of Sponsor. The Principal Investigator further agrees to provide thirty (30) days prior to submission for publication or presentation to Sponsor to review copies of abstracts or manuscripts for publication (including texts of oral presentations) which report any results of the Protocol study.